CLINICAL TRIAL: NCT06275230
Title: Establishment of Human Lung Stem Cell Proliferation System and Organoid Construction in Chronic Obstructive Pulmonary Disease
Brief Title: Establishment of Human Lung Stem Cell Proliferation System and Organoid Construction in COPD
Status: Recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Principal Investigator, China-Japan Friendship Hospital
Other Study IDs: ZRJY2021-BJ08-02-07
Record Dates: First submitted 2024-02-17; First posted 2024-02-23 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; organoid; human lung stem cells
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- chronic obstructive pulmonary disease: Patients with COPD undergoing bronchoscope.

SUMMARY:
The goal of this study is to proliferate human lung stem cell in vitro in order to establish a lung organoid derived from patients with COPD. The main question it aims to answer are:

* Can human lung stem cell proliferate in vitro.
* Can a lung organoid derived from patients with COPD be established. Participants will be sampled during pulmonary bronchoscope for organoid establishment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age under 55, regardless of gender
* 2. Patients with COPD lung disease who are going to undergo bronchoscopic biopsy
* 3. No genetic diseases and other respiratory diseases

Exclusion Criteria:

* Other conditions determined by the investigators to be unsuitable for inclusion, such as difficult sampling, difficult follow-up, and complicated with other serious diseases

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: COPD Patients with indications of bronchoscopic biopsy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Patients completed bronchoscope. | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China